CLINICAL TRIAL: NCT06360887
Title: Management of Proximal Humerus Fractures in Elderlies: a Clinical Trial
Brief Title: Management of Proximal Humerus Fractures in Adults: a Clinical Trial
Status: Not yet recruiting | Type: Observational
Sponsor: Regional Hospital of Bolzano (Other)
Responsible Party: Principal Investigator, Malte Nikolas Witte, Medical Doctor, Regional Hospital of Bolzano
Other Study IDs: DRKS00030614
Record Dates: First submitted 2024-03-28; First posted 2024-04-11 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Shoulder Fractures
MeSH Terms: conditions — Shoulder Fractures | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Conservative: Participants allocated to conservative management will receive an orthosis (Gilchrist) for a minimum of four weeks. Using Gilchrist, the upper arm of the injured side is secured in abduction and internal rotation with the weight of the arm held by a ring around the patient's neck. At four weeks, plain radiographs of the shoulder will be conducted to ascertain the presence of the bony callous. If a bony callous is not present, the patient will maintain Gilchrist and plain radiographs of the shoulder will be conducted on a biweekly basis until a bony callous will be evident. If a bony callous is present, the patient will start a structured program of rehabilitation.
  Interventions: Procedure: Conservative
- Open Reduction Internal Fixation: Participants allocated to ORIF will undergo surgery within 72 hours from the diagnosis using a standard deltopectoral approach. An angular stable plate is used in all patients following manufacturer instructions. No drains will be used.
  Interventions: Procedure: ORIF
- Closed Reduction Percutaneous Pinning: Participants allocated to CRPP will be positioned in a beach chair under total anesthesia. The fracture is repositioned under fluoroscopic guidance using manual traction. The osteosynthesis is then done using Kirschner wires.The arm is placed into a Gilchrist for four weeks. At four weeks, plain radiographs of the shoulder will be conducted to ascertain the presence of the bony callous. If a bony callous is not present, the patient will maintain Gilchrist and plain radiographs of the shoulder will be conducted on a biweekly basis until a bony callous will be evident. If a bony callous is present, the Kirschner wires will be removed and the patient will start a structured program of rehabilitation.
  Interventions: Procedure: CRPP

INTERVENTIONS:
Procedure: Conservative — Conservative treatment
  Groups: Conservative
Procedure: ORIF — Open surgery
  Groups: Open Reduction Internal Fixation
Procedure: CRPP — Minimal invasive surgery
  Groups: Closed Reduction Percutaneous Pinning

SUMMARY:
Prospective patient registry examining the outcome of three different treatment methods for proximal humerus fractures in elderlies: conservative treatment, open and minimal invasive surgical treatment.

DETAILED DESCRIPTION:
The present study shall be conducted in accordance with the SPIRIT 2013 statement: defining standard protocol items for clinical trials. All patients who sustained a PHF and presented at the Department of Orthopedics at the Academic Hospital of Bolzano (Italy) will be prospectively incited to participate in the present clinical trial. Patient recruitment will begin in April 2024, and end in April 2026. The follow-up period will start in October 2024, and end in April 2028. Data analysis will commence in October 2024 and end in April 2028. The present study shall be conducted according to the principles of the Declaration of Helsinki. The authors receive no financial support for the research, authorship, and/or publication of this article. The protocol of the study has been prospectively registered and approved by the German Registry of Clinical Trials (ID DRKS00030614). Ethics approval has been received from the Ethic Committee of the South Tyrolean Health Authority, Bolzano, Italy (ID 2022374 of June 22, 2023). All surgical and conservative procedures under analysis are already routinely carried out at the Department of Orthopaedics and Trauma Surgery of the Academic Hospital of Bolzano, Italy. Patients who meet the inclusion criteria and agree to participate in the study by signing the consent form and the personal data processing form will be included in the study.

Data curation Personal data, including sensitive data, will be pseudonymised and associated with a code from which it will be impossible to trace the patient's identity. Only the Principal Investigator and sub-investigators of the study will be able to link the code to the name. The pseudonymised data will be collected in a table of Microsoft Office Excel version 16 (Microsoft Corporation, Redmond, US).

Statistical analyses Assuming an actual difference in means between the test and reference group of 3 units and a pooled standard deviation of 5 units, the study would require a sample size of 117 patients for each group (i.e. a total sample size of 351, assuming equal group size), to obtain a power of 80% and a significance level of 5%, to declare the superiority of a technique with a margin of prominence of 5 units, assuming a minimum clinically important difference OSS of 2.7/100 .

ELIGIBILITY:
Inclusion Criteria:

1. adults who sustained a Proximal Humerus Fracture within the last week
2. type of Proximal Humerus Fracture AO 11-(A2, A3), 11- (B1, B2, B3)
3. BMI lower than 40 Kg/m2

Exclusion Criteria:

1. stress fractures
2. revision setting
3. open fractures
4. fractures associated with a neurologic lesion; previous fractures or bony procedure at the homolateral side
5. patients unable to understand the procedure or instructions for rehabilitation
6. terminal patients
7. patients presenting multiple injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults presenting at our hospital with proximal humerus fractures that meet the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 351 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Oxford Shoulder Score | 6, 12, and 24 months after surgery
  The primary endpoint of interest will be the Oxford Shoulder Score. The Oxford Shoulder Score is a patient-reported outcome measure developed to evaluate perceived pain and quality of life in subjects who received a shoulder operation. It can be used independently from the performed surgical treatment, excluding only surgical stabilisations. As the Italian province of Bolzano is bilingual (Italian and German), the Italian and German versions of the Oxford Shoulder Score shall be administered. Both versions of the Oxford Shoulder Score are valid and reliable, with high internal consistency and reproducibility. The Oxford Shoulder Score comprises 12 items with five possible answers each: pain (four items) and quality of life (eight items).
  The Oxford Shoulder Score contains two subscales, pain (20 points) and activities of daily living (40 points). Scores range from 0 to 60, with a higher score being consistent with increased disability.

SECONDARY OUTCOMES:
The visual analogue scale | 6, 12, and 24 months after surgery
  The visual analogue scale (VAS) is a scale used to determine the pain intensity. The minimum value is 0, the maximum value is 10, with 0 meaning no pain and 10 the worst pain imaginable.
Rate of complications | 6, 12, and 24 months after surgery
  persistent pain, frozen shoulder, malunion, surgery, nerve damage

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Migliorini, Dr., Principal Investigator — employee
Locations (1):
- Academic Hospital of Bolzano (SABES-ASDAA), Bolzano, Trentino-Alto Adige, Italy

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: when data is publicised
Access Criteria: information will be shared if asked for with other researchers